CLINICAL TRIAL: NCT06861894
Title: Active Surveillance After Neoadjuvant Adebrelimab Combined With Chemoradiotherapy for Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Active Surveillance After Neoadjuvant Adebrelimab Combined With Chemoradiotherapy for Resectable ESCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhigang Li (Other)
Responsible Party: Sponsor-Investigator, Zhigang Li, Chief of Department of Esophageal Surgery, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-EC-II-017
Record Dates: First submitted 2025-03-03; First posted 2025-03-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — 130-nm albumin-bound paclitaxel; Carboplatin; Radiation; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- perioperative treatment with adebrelimab and CRT (Experimental)
  Interventions: Drug: Adebrelimab and nab-paclitaxel and carboplatin; Radiation: Radiation; Procedure: standard oesophagectomy; Other: active surveillance

INTERVENTIONS:
Drug: Adebrelimab and nab-paclitaxel and carboplatin — Adebrelimab combined with nab-paclitaxel and carboplatin as neoadjuvant therapy
Radiation: Radiation — concurrent chemoradiotherapy
Procedure: standard oesophagectomy — standard oesophagectomy
Other: active surveillance — active surveillance

SUMMARY:
In this prospective trial, patients demonstrating clinical complete response (cCR) as determined by a standard response assessment protocol (incorporating clinical and molecular diagnostic methods) will be offered organ-sparing management following neoadjuvant therapy with adebrelimab (anti-PD-L1) concurrent with chemoradiotherapy. The primary endpoint is 2-year overall survival rate in this watch-and-wait cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects signed the informed consent and volunteered to participate in the study.
2. Esophageal squamous cell carcinoma confirmed by histology or cytology.
3. Thoracic esophageal squamous cell carcinoma confirmed by CT or pet-CT, which is classified as cII-III (AJCC 8th).
4. Expect to have R0 resection
5. In age from 18 to 75.
6. ECOG PS: 0~1.
7. Have not received any anti-tumor treatment for esophageal cancer in the past, including radiotherapy, chemotherapy, surgery, etc.
8. No contraindications to surgery.
9. Has sufficient organ function including (1) Blood routine: NE≥1.5×109/L; PLT≥100×109/L; HGB≥90 g/L (2)Comprehensive Metabolic Panel: bilirubin≤ 1.5×ULN; ALT≤2.5×ULN; AST≤2.5×ULN; sCr≤1.5×ULN or CrCl≥50 mL/min（Cocheroft-Gault) (3) Coagulation function: INR≤1.5; APTT≤1.5×ULN
10. Women of childbearing age must undergo a serological pregnancy test within 72 hrs before first administration. Women of childbearing age, or male subjects with childbearing age female partners, must take contraceptive measures from the first dose to three months after last administration.
11. Good compliance, willing to comply with follow-up schedules.

Exclusion Criteria:

1. Subjects have received or are receiving any of:

   1. anti-tumor interventions such as radiotherapy, chemotherapy, or other medications.
   2. immunosuppressants or systemic glucosteroids (prednisone equivalence> 10mg/d) within 2 weeks before the first administration, inhaled or topical use of glucosteroids (prednisone equivalence>10mg/d) is allowed if no known active autoimmune disease.
   3. live vaccine within 4 weeks before the first administration.
   4. major surgery or major injury within 4 weeks before the first administration.
2. Cancer-related exclusion criteria

   1. other cancers instead of ESCC
   2. unresectable or metastatic ESCC
   3. not comply with cⅡ-Ⅲ（cT2N1-2M0 or cT3N0-2M0, AJCC 8th）
   4. Subjects with other malignant tumors within 5 years before the first administration, but subjects with cervical carcinoma in situ, skin basal cell carcinoma, skin squamous cell carcinoma, localized prostate cancer received radical surgery and ductal carcinoma in situ that have received radical treatment and do not need other treatment can be included)
3. Other criteria

   1. Subjects have uncontrolled cardiovascular diseases, such as 1) heart failure ≥ NYHA class 2, 2) unstable angina 3) myocardial infarction within 1 year; 4) supraventricular or ventricular arrhythmia that needs treatment
   2. Subjects with any known active autoimmune disease
   3. Pregnant or breastfeeding female
   4. Presence of allergy or hypersensitivity to investigational medications
   5. HIV-positive or active hepatitis B (HBsAg positive and HBV-DNA ≥2000 IU/ml or ≥ 104 copies/mL) or active hepatitis C (HCV antibody positive) or active tuberculosis
   6. Investigators assessed there might be other factors that cause subjects to withdraw.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
2-year OS rate | 24 months
  An overall survival (OS) is defined as the time from treatment to death, regardless of disease recurrence.

SECONDARY OUTCOMES:
cCR rate | 12 months
  A clinical complete response rate (cCR) is defined as the complete disappearance of tumor lesions.
median EFS | 24 months
  An event-free survival (EFS) is defined as the duration from the start of treatment until disease recurrence or death from any cause, whichever occurs first.
median OS | 24 months
  An overall survival (OS) is defined as the time from treatment to death, regardless of disease recurrence.
Incidence, type and severity of adverse events as assessed by CTCAE 5.0 | 24 months
  Including adverse events and complications. Incidence of adverse events using CTCAE 5.0; grade 3 adverse events and higher-grade will be reported.
quality of life (QOL) | 24 months
  Evaluate quality of life using EORTC QLQ-C30
quality of life (QOL) assessed by EORTC QLQ-OES18 | 24 months
  Evaluate quality of life using EORTC QLQ-OES18

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided